CLINICAL TRIAL: NCT00734682
Title: A Phase I Trial of Nanoliposomal CPT-11 (NL CPT-11) in Patients With Recurrent High-Grade Gliomas
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Principal Investigator, Michael Prados, Professor, University of California, San Francisco
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08103; NCT00745082 (obsolete NCT alias)
Record Dates: First submitted 2008-08-13; First posted 2008-08-14 (Estimated); Last update posted 2015-01-07 (Estimated); Status verified 2014-12

CONDITIONS: Glioblastoma; Gliosarcoma; Anaplastic Astrocytoma; Anaplastic Oligodendroglioma
Keywords: Glioblastoma; Gliosarcoma; Anaplastic Astrocytoma; Anaplastic Oligodendroglioma; Anaplastic Mixed Oligoastrocytoma; Malignant Astrocytoma NOS; Nanoliposomal CPT-11; liposomal irinotecan
MeSH Terms: conditions — Glioblastoma; Gliosarcoma; Astrocytoma; Oligodendroglioma | interventions — irinotecan sucrosofate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Nanoliposomal CPT-11 (Experimental): All patients are treated with nanoliposomal CPT-11
  Interventions: Drug: Nanoliposomal CPT-11

INTERVENTIONS:
Drug: Nanoliposomal CPT-11 — Depending on UGT1A1 genotyping status, patients are either given a starting dose of 120 mg/m^2 (wild type) or 60 mg/m^2 IV q3 weeks.
  Other Names: NL CPT-11; liposomal irinotecan

SUMMARY:
This is a Phase I study of Nanoliposomal CPT-11 in patients with Recurrent high-grade gliomas. Patients must have a histologically proven intracranial malignant glioma, which includes glioblastoma multiforme (GBM), gliosarcoma (GS), anaplastic astrocytoma (AA), anaplastic oligodendroglioma (AO), anaplastic mixed oligoastrocytoma (AMO), or malignant astrocytoma NOS (not otherwise specified). Patients who are wild type or heterozygous for the UGT1A1*28 gene will received Nanoliposomal CPT-11. The total anticipated accrual will be approximately 36 patients (depending upon the actual MTD). The investigators hypothesis is that this new formulation of CPT-11 will increase survival over that seen in historical controls who have recurrent gliomas because CPT-11 will be encapsulated in a liposome nanoparticle, which has been seen to reduce toxicities from the drug.

DETAILED DESCRIPTION:
Patients with recurrent malignant glioma will receive Nanoliposomal CPT-11 at the time of relapse. The dose will be adjusted according to a phase-1 dose escalation scheme. Patients will receive drug intravenously every 3 weeks until tumor progression or excessive toxicity. Weekly follow up will occur to assess toxicities during the DLT phase of the trial. Patients will have different dose escalation if UGT1A1 is 6/6 versus UGT1A1 is 6/7. Patients with UGT 1A1 of 7/7 will not be eligible. All patients must have UGT 1A1 status know as an eligibility requirement. Patients will be followed for both toxicity and progression, and progression will be evaluated by MR imaging every 6 weeks. Pharmacokinetics will be obtained in the first treatment cycle.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically proven intracranial malignant glioma are eligible . -All patients must sign an informed consent

  * Patients must be > 18 years old, and with a life expectancy > 8 weeks.
  * Patients must have a Karnofsky performance status of > 60.
* Patients must have recovered from the toxic effects of prior therapy
* Patients must have adequate bone marrow function (WBC > 3,000/µl, ANC > 1,500/mm3, platelet count of > 100,000/mm3, and hemoglobin > 10 gm/dl), adequate liver function (SGOT and bilirubin < 2 times ULN), and adequate renal function (creatinine < 1.5 mg/dL and/or creatinine clearance > 60 cc/min) Patients must have shown radiographic evidence for tumor progression by MRI or CT scan. A scan should be performed within 14 days prior to registration and on a steroid dose that has been stable for at least 5 days. -Patients having undergone recent resection of recurrent or progressive tumor will be eligible as long as all of the following conditions apply:

  * They have recovered from the effects of surgery.
  * Residual disease following resection of recurrent malignant glioma is not mandated for eligibility into the study.
* Patients must have failed prior radiation therapy
* Patients with prior therapy that included interstitial brachytherapy or stereotactic radiosurgery must have confirmation of true progressive disease
* Women of childbearing potential must have a negative ß-HCG pregnancy test documented within 14 days prior to registration.
* Patients may have had treatment for any number of prior relapses.

Exclusion Criteria:

* Patients must not have any significant medical illnesses that in the investigator opinion cannot be adequately controlled
* Patients with a history of any other cancer (except non-melanoma skin cancer or carcinoma in-situ of the cervix), unless in complete remission and off of all therapy for that disease for a minimum of 3 years are ineligible.
* Patients must not have active infection or serious intercurrent medical illness.
* Patients must not be pregnant/breast feeding and must agree to practice adequate contraception.
* Patients must not have any disease that will obscure toxicity or dangerously alter drug metabolism.
* Patients must not have received prior therapy with irinotecan.
* Patients with 7/7 (homozygous) UGT1A1*28 genotyping will be excluded from the study.
* Patients receiving enzyme-inducing anticonvulsants or other enzyme inducing drugs are excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2008-08; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
To assess the safety and pharmacokinetics of NL CPT-11 in patients with recurrent malignant glioma stratified based on UGT1A1 genotyping. | 1-2 years

SECONDARY OUTCOMES:
To determine the maximum tolerated dose of NL CPT-11 in these patient populations. | 1-2 years

CONTACTS AND LOCATIONS:
Overall Officials: Michael Prados, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States